CLINICAL TRIAL: NCT02337374
Title: Do Urodynamics Superior to 25 Years of Clinical Expertise Predict Mid-Urethral Sling Failure?
Brief Title: Predictive Role of Urodynamics on Mid-urethral Sling Failure
Acronym: UPMUSF
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, serdar aydin, MD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSSRTH2010-06
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urodynamics; Midurethral sling; Transobturator tape (TOT); Tension free vaginal tape (TVT)
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Midurethral sling mesh

SUMMARY:
Purpose The aim of this study is to investigate the contribution of preoperative urodynamics to mid-urethral slings (MUS) success for developing an algorithm that uses conventional and easily accessible tools Methods Women with stress urinary incontinence and who desired surgical correction of their incontinence were included in the study. The selection of the procedure was according to an algorithm used in an institution developed by a chief of urogynecology department who had 25 years of urogynecology experience. Urodynamic and baseline factors that may be associated with surgery failure were analyzed in MUS failure.

ELIGIBILITY:
Inclusion Criteria:

* Documented pure or predominant SUI symptoms for at least 3 months, along with a positive standardized urinary stress test

Exclusion Criteria:

* prior incontinence surgery, post-void residual volumes of greater than 100 ml, a history of chronic inguinal or vulvar abscess, hidradenitis suppurativa, genitourinary fistula or urethral diverticulum, reversible cause of incontinence (i.e., drug effect), or any contraindication to surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with stress urinary incontinence and who desired surgical correction of their incontinence
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Mid urethral sling surgery failure | after june 2010